CLINICAL TRIAL: NCT02345395
Title: Safety Study of Minimally Invasive Approaches to Unruptured Anterior Circulation Aneurysms
Acronym: MININCRUSP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TRANSPALPEBRAL USP
Record Dates: First submitted 2015-01-19; First posted 2015-01-26 (Estimated); Last update posted 2015-01-26 (Estimated); Status verified 2014-01

CONDITIONS: Cerebral Aneurysm; Aneurysm, Middle Cerebral Artery; Aneurysm, Anterior Communicating Artery; Aneurysm, Posterior Communicating Artery; Aneurysm, Carotid Artery; Brain Aneurysm
Keywords: Brain Aneurysm; Pterional Craniotomy; MiniPterional Craniotomy; Transpalpebral Approach; Unruptured Brain Aneurysm
MeSH Terms: conditions — Intracranial Aneurysm; Aneurysm

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Transpalpebral Approach (Experimental): Aneurysm Clipping - Patients will be submitted to a Transpalpebral Approach to Unruptured Anterior Circulation Aneurysm and they will be discharged from the hospital on the next day.
  Interventions: Procedure: Aneurysm Clipping
- NanoPterional Approach (Experimental): Aneurysm Clipping - Patients will be submitted to a Modified MiniPterional Approach (Nanopterional) to Unruptured Anterior Circulation Aneurysm and they will be discharged from the hospital on the next day.
  Interventions: Procedure: Aneurysm Clipping
- Classical Pterional Craniotomy (Sham Comparator): Aneurysm Clipping - Patients will be submitted to a Classical Pterional Approach to Unruptured Anterior Circulation Aneurysm and they will be discharged from the hospital 4-5 days after the procedure.
  Interventions: Procedure: Aneurysm Clipping

INTERVENTIONS:
Procedure: Aneurysm Clipping — All Patients will be submitted to a surgical intervention in order to clip their unruptured brain aneurysm

SUMMARY:
The study is designed to evaluate the efficacy and safety of minimally invasive neurosurgical techniques for patients with incidental cerebral aneurysms of the anterior circulation in the Hospital das Clínicas of the University of São Paulo Medical School.

DETAILED DESCRIPTION:
Minimally Invasive Neurosurgery is a inexorable tendency and it is already a reality in many centers of the world. It is a broad and relative concept and there is few consistent medical data to validate its benefits. In this manner, this is the first clinical trial in Brazil questioning the safety of the of minimally invasive surgery to treat incidental cerebral aneurysms of the anterior circulation. For countries like Brazil, the indirect demonstration of reduction in hospital costs through lower hospital stays is a breakthrough to provide better health for the entire population.

Patients with the diagnosis of incidental brain aneurysms of the anterior circulation will be recruited from the spontaneous demand of the Hospital das Clínicas of University of São Paulo Medical School. The investigators expect to recruit 60 patients for the experimental group and 60 for the control group.

In the study group patients will be submitted to a minimally invasive approach (transpalpebral mini fronto-orbital craniotomy or modified minipterional craniotomy). All patients in this group will be submitted to surgery starting at 8 o'clock in the morning. After 6 hours of the end of surgery, all patients will have a control CT scan and if the result is adequate, they are going to be discharged from the ICU with no IV drugs. The hospital discharge will be in the next day. The control group are patients that will be submitted to a classical pterional craniotomy with hospital discharge occurring in 4-5 days.

All patients will be submitted to the standard care offered by the Hospital das Clinicas. All surgical and ambulatory data will be collected by the main investigators (Dr. Mauricio Mandel and Dr. Eberval Figueiredo). The adverse events will be promptly reported to the chair of the department and to the CAPPESQ (the ethics committee of the hospital).

Ambulatory data will be collected during the regular post operative medical appointments and a web based questionnaire. The post operative follow-up is unified in only one ambulatory center and day (thursdays mornings).

Statistical analysis will compare primary and secondary objectives of the two groups, as specified in the study protocol.

ELIGIBILITY:
Inclusion Criteria:

* Patients with the diagnosis of incidental unruptured cerebral aneurysms (4mm to 2cm)

Exclusion Criteria:

* Patients who do not have adequate family care during the immediate post-operative period (the patient's family must commit to stay with the patient in the first five days after hospital discharge)
* Patients who are unable to communicate by telephone
* People with cardiovascular disease, liver or kidney failure.
* Pregnant women or breastfeeding
* Patients with coagulation abnormalities
* Patients with High Surgical Risk evaluated by different risk scores (ASA, AHA, Goldman, Detsky)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2013-09; Primary Completion 2015-07 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Effective Aneurysm Clipping (no residual cerebral aneurysm) | 3 months after surgery
  All patients will be submitted to a post operative angiography to asses the presence of residual cerebral aneurysm after clipping.

SECONDARY OUTCOMES:
All Cause Mortality | 1 year
Neurological Outcome | 1 year
  All patients will be classified with the Glasgow Outcome Scale, Rankin Scale
Cosmetic Outcome | 1 year
  Comparison of pre and post operative photos and asses of patients satisfaction
Surgical Safety assessed by number and description of Surgical Complications (infection rate, postoperative epidural/ contusional hematomas, number of reoperations, need of blood transfusion) | 1 year
Early Hospital Discharge | 15 days
  Safety of early Discharge in the Experimental Groups (need of early hospital readmission? and its causes)

OTHER OUTCOMES:
Quality of Life | 15 days, 3 months, 6 months and 1 year
  Whoqol-bref questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Eberval G Figueiredo, MD, PhD, Study Director — University of Sao Paulo
Locations (1):
- Hospital das Clínicas of University of São Paulo Medical School, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Ohjimi H, Taniguchi Y, Tanahashi S, Era K, Fukushima T. Accessing the Orbital Roof via an Eyelid Incision: The Transpalpebral Approach. Skull Base Surg. 2000;10(4):211-6. doi: 10.1055/s-2000-9337. PMID 17171150
- [Background] Andaluz N, Romano A, Reddy LV, Zuccarello M. Eyelid approach to the anterior cranial base. J Neurosurg. 2008 Aug;109(2):341-6. doi: 10.3171/JNS/2008/109/8/0341. PMID 18671651
- [Background] Abdel Aziz KM, Bhatia S, Tantawy MH, Sekula R, Keller JT, Froelich S, Happ E. Minimally invasive transpalpebral "eyelid" approach to the anterior cranial base. Neurosurgery. 2011 Dec;69(2 Suppl Operative):ons195-206; discussion 206-7. doi: 10.1227/NEU.0b013e31821c3ea3. PMID 21499147
- [Background] Figueiredo EG, Deshmukh V, Nakaji P, Deshmukh P, Crusius MU, Crawford N, Spetzler RF, Preul MC. An anatomical evaluation of the mini-supraorbital approach and comparison with standard craniotomies. Neurosurgery. 2006 Oct;59(4 Suppl 2):ONS212-20; discussion ONS220. doi: 10.1227/01.NEU.0000223365.55701.F2. PMID 17041490
- [Background] Figueiredo EG, Deshmukh P, Nakaji P, Crusius MU, Crawford N, Spetzler RF, Preul MC. The minipterional craniotomy: technical description and anatomic assessment. Neurosurgery. 2007 Nov;61(5 Suppl 2):256-64; discussion 264-5. doi: 10.1227/01.neu.0000303978.11752.45. PMID 18091240